CLINICAL TRIAL: NCT06587009
Title: Director of Rehabilitation Medicine
Brief Title: Application of Shock Wave Technique in Conservative Treatment of Rotator Cuff Tear
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2024208
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Rotator Cuff Tear
Keywords: Shock wave technique; Conservative treatment
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESWT group (Experimental): Patients who receive shock wave technique
  Interventions: Procedure: Shock wave therapy
- Control group (Experimental): Patients who receive conventional conservative treatment
  Interventions: Procedure: Conventional conservative treatment

INTERVENTIONS:
Procedure: Shock wave therapy — Received shock wave therapy 7 times a week and functional exercise therapy intervention
  Arms: ESWT group
Procedure: Conventional conservative treatment — Conventional conservative treatment and functional exercise were given
  Arms: Control group

SUMMARY:
This study is a prospective cohort study and is a single-center clinical trial. Sample: This study will enroll about 22 patients from the Department of Sports Medicine and rehabilitation outpatient department of Beijing Third Hospital who are diagnosed with rotator cuff tear and choose conservative treatment.

DETAILED DESCRIPTION:
A single-center randomized controlled clinical trial was conducted to compare the effect of ESWT combined with conventional rehabilitation training on patients with rotator cuff tear. To explore the effect of ESWT on the clinical efficacy of patients with rotator cuff tear, and to explore the application of shockwave technology in the conservative treatment of rotator cuff tear. It provides a new treatment idea for patients with rotator cuff tear who choose conservative treatment, promotes tendon healing for patients with partial rotator cuff tear, improves shoulder joint function, and provides a new treatment plan for patients to accelerate their return to life and exercise, and provides a theoretical basis for the clinical application of ESWT.

ELIGIBILITY:
Inclusion Criteria:

* Identify patients with rotator cuff tears and choose conservative treatment
* Able to complete cardiopulmonary exercise tests
* Able to cooperate with rehabilitation training and complete questionnaire survey

Exclusion Criteria:

* Previous shoulder surgery history
* Irreparable rotator cuff damage
* Retear after ARCR

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
pain VAS score | 6 weeks, 3 months, and 6 months after surgery
  pain levels in patients, ranging from 0 to 10, with a higher score indicating more intense pain.
ASES score | 6 weeks, 3 months, and 6 months after surgery
  The American Shoulder and Elbow Surgeons (ASES) score is the most commonly used score to describe the function of patients' shoulder joints, ranging from 0 to 100. The higher the score, the better the function of patients' shoulder joints.
MRI evaluation | 3 months and 6 month after surgery
  Through MRI qualitative and quantitative analysis, evaluate the tendon healing status after rotator cuff repair surgery.
UCLA score | 6 weeks, 3 months and 6 months after surgery
  The UCLA Shoulder Score combines input from both the physician and the patient and totals range from 0 to 35, 0s indicating worse shoulder function and 35s indicating better shoulder function outcomes.

SECONDARY OUTCOMES:
Active shoulder ranges of motion | 6 weeks, 3 months, and 6 months after surgery
  internal rotation at the side, and external and internal rotation at 90° of abduction

CONTACTS AND LOCATIONS:
Overall Officials: Guoqing Cui, Study Chair — Peking University Third Hospital
Locations (1):
- PekingUTH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No